CLINICAL TRIAL: NCT06530407
Title: Gender-Based Comparison of the Immediate Effects of Lower Extremity Static Stretching Exercises on Vertical Jump in Sedentary Individuals
Brief Title: Comparison of the Immediate Effects of Lower Extremity Static Stretching Exercises on Vertical Jump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Duygu Şahin Altaç, PT, MSc., Halic University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28.07.2024-İEU
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Stretch
Keywords: strech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 10 sedentary women
  Interventions: Other: Static streching exercise
- Group 2 (Experimental): 10 sedentary men
  Interventions: Other: Static streching exercise

INTERVENTIONS:
Other: Static streching exercise — Static stretching exercises were applied to the M. Gastrocnemious and M. Hamstring muscle groups for both groups. The exercises were applied as a set, with three repetitions for 15 seconds on each leg, with a 20-second rest between repetitions. Static stretching was applied by slowly stretching the relevant muscle group to the point of sensitivity, without straining the pain threshold, and waiting in that position. All stretching exercises lasted an average of 6 minutes.

SUMMARY:
The aim of this study is to compare the immediate effects of lower extremity static stretching exercises on vertical jump in sedentary individuals based on gender.

DETAILED DESCRIPTION:
The study was conducted on 10 female (Group 1) and 10 male (Group 2) university students. The vertical jump height (VJH) of the individuals who agreed to participate in the study was measured with a wireless jumping platform. After the initial evaluations, lower extremity static stretching exercises targeting the M. Gastrocnemious and M. Hamstring muscles were applied to the participants in both groups. The VJH of the participants was re-evaluated immediately after the application. Both pre-post evaluations and female-male comparison evaluations will be performed for the statistical analysis of the data.Statistical analysis will be performed with SPSS 24.0 program. If the data is parametric, paired sample t-test will be used for within-group evaluation; independent sample t-test will be used for between-group evaluation. If the data is non-parametric, Wilson test will be used for within-group evaluation and Mann Whitney U test will be used for between-group evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 18-25

Exclusion Criteria:

* Having balance problems for any reason
* Having a history of lower extremity surgery
* Having a musculoskeletal problem within the last year
* Doing regular exercise within the last year

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Group 1: 10 sedantary women Group 2: 10 sedantary men
Enrollment: 20 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Vertical jump height | at baseline and immediately after the lower extremity static stretching exercise program
  DSY was measured with a wireless jumping platform (Ezejump, Australia). Participants were subjected to three squat jump tests on this platform with free intervals between repetitions and the maximum value obtained from the test was recorded as the vertical jump height.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Şahin Altaç, PT, MSc., Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marek SM, Cramer JT, Fincher AL, Massey LL, Dangelmaier SM, Purkayastha S, Fitz KA, Culbertson JY. Acute Effects of Static and Proprioceptive Neuromuscular Facilitation Stretching on Muscle Strength and Power Output. J Athl Train. 2005 Jun;40(2):94-103. PMID 15970955
- [Result] Dalrymple KJ, Davis SE, Dwyer GB, Moir GL. Effect of static and dynamic stretching on vertical jump performance in collegiate women volleyball players. J Strength Cond Res. 2010 Jan;24(1):149-55. doi: 10.1519/JSC.0b013e3181b29614. PMID 20042927
- [Result] Markovic G, Dizdar D, Jukic I, Cardinale M. Reliability and factorial validity of squat and countermovement jump tests. J Strength Cond Res. 2004 Aug;18(3):551-5. doi: 10.1519/1533-4287(2004)182.0.CO;2. PMID 15320660